CLINICAL TRIAL: NCT04074421
Title: Effects of Continuous Treatment With Rifaximin and Probiotics on the Gut Microbiota of Patients With Diarrhoea-predominant Irritable Bowel syndrome-a Multicentre Controlled Study
Brief Title: Effects of Continuous Treatment With Rifaximin and Probiotics on the Gut Microbiota of Patients With IBS-D
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); RenJi Hospital (Other); Peking Union Medical College Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); The Central Hospital of Lishui City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: (2019) Study No. 413
Record Dates: First submitted 2019-08-26; First posted 2019-08-30 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2019-08

CONDITIONS: IBS - Irritable Bowel Syndrome; Gut Microbiota
Keywords: Rifaximin; Probiotics; IBS-D; gut microbiota
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rifaximin group (Active Comparator): Repeating treatment of Rifaximin
  Interventions: Drug: Rifaximin
- Probiotics group (Sham Comparator): Sequential treatment of probiotics called Bacillus subtilis and Enterococcus faecium
  Interventions: Drug: Probiotic Formula
- Placebo group (Placebo Comparator): Placebo control group
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Rifaximin — A non-aminoglycoside intestinal antibiotic, 400mg, twice one day for 2 weeks.
  Arms: Rifaximin group
Drug: Probiotic Formula — A probiotic called Enterococcus faecium, 500mg, triple one day for 4 weeks.
  Other Names: probiotic formula Bacillus subtilis and Enterococcus faecium
  Arms: Probiotics group
Drug: Placebo oral tablet — Placebo oral tablet that has no therapeutic effect
  Other Names: Placebo
  Arms: Placebo group

SUMMARY:
We will use the latest Rome IV criteria to recruit IBS-D patients and evaluate the effects of repeated treatment with rifaximin and sequential treatment with rifaximin and probiotics on different symptoms and quality of life. High-throughput sequencing combined with real-time quantitative PCR will be used to comprehensively analyze the effects of different drugs on intestinal flora. The study has important guiding significance for the treatment of patients with IBS-D.

DETAILED DESCRIPTION:
According to the Rome IV diagnostic criteria, 200 patients with with diarrhoea-predominant irritable bowel syndrome (IBS-D) from the multi-center (8 units in the country) will be enrolled. The IBS Severity Inventory (IBS-SSS) and IBS Quality of Life Scores (QOL) will be used to evaluate the effect of treatments. Retreatment patients who are initially treated and not satisfied with the improvement of symptoms and quality of life will be treated with Rifaximin for 2 weeks. Fecal specimens will be collected from patients who responded to treatment, and the fecal bacteria will be analyzed by real-time polymerase chain reaction (PCR) using 16 S ribosomal ribonucleic acid (rRNA) gene. Patients who responded to Rifaximin treatment will be randomized into A (Probiotics group) and B (Placebo group). IBS symptom grade score and quality of life score will be evaluated before and after treatment, and fecal specimens of the responding patients will be collected for intestinal probiotics and harmful bacteria detection.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old;
* in line with the diagnostic criteria of diarrhea-type irritable bowel syndrome Roman IV；
* blood routine, blood biochemistry, stool examination and colonoscopy within 2 years are no problem;
* no intestinal warning symptoms

Exclusion Criteria:

* suffering from severe heart, lung, liver, kidney, nervous system diseases;
* suffering from mental disorders caused by schizophrenia, brain organic and physical diseases;
* suffering from other diseases that may affect intestinal function (such as diabetes, thyroid disease);
* History of previous abdominal surgery (excluding history of cholecystectomy or appendectomy);
* pregnant or lactating women;
* have undergone colonoscopy in the past month or accept other bowel preparation operations;
* In the past 1 month, have used antibiotics, antidiarrheal agents, intestinal flora regulation, Chinese medicine and other drugs;
* have participated in other dietary treatments;
* understand communication barriers, unable to communicate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-05-10 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
the IBS symptom grade score | baseline
  The IBS Severity Inventory (IBS-SSS) will be used to evaluate the IBS symptom grade score The IBS Severity Inventory (IBS-SSS) will be used to evaluate the IBS symptom grade score
the quality of life score | baseline
  IBS Quality of Life Scores (QOL) will be used to evaluate the quality of life score
the IBS symptom grade score | 2 weeks
  The IBS Severity Inventory (IBS-SSS) will be used to evaluate the IBS symptom grade score The IBS Severity Inventory (IBS-SSS) will be used to evaluate the IBS symptom grade score
the quality of life score | 2 weeks
  IBS Quality of Life Scores (QOL) will be used to evaluate the quality of life score
the IBS symptom grade score | 12 weeks
  The IBS Severity Inventory (IBS-SSS) will be used to evaluate the IBS symptom grade score
the quality of life score | 12 weeks
  IBS Quality of Life Scores (QOL) will be used to evaluate the quality of life score
16 S rRNA (ribosomal ribonucleic acid) to detect gut microbiota | 12 weeks
  16 S rRNA (ribosomal ribonucleic acid) sequencing will be applied to determine the change of microbial community
16 S rRNA (ribosomal ribonucleic acid) to detect gut microbiota | baseline
  16 S rRNA (ribosomal ribonucleic acid) sequencing will be applied to determine the change of microbial community
16 S rRNA (ribosomal ribonucleic acid) to detect gut microbiota | 2 weeks
  16 S rRNA (ribosomal ribonucleic acid) sequencing will be applied to determine the change of microbial community

CONTACTS AND LOCATIONS:
Overall Officials: Liangjing Wang, Ph.D, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
The study is not yet recruiting and unfinished.